CLINICAL TRIAL: NCT07308119
Title: Comparison Between Pilates Exercises and Aerobic Exercises in Primary Dysmenorrhea
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rana Salem Abdelghany Ali (Other)
Responsible Party: Sponsor-Investigator, Rana Salem Abdelghany Ali, Principal Investigator, Kafrelsheikh University
Organization: Kafrelsheikh University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-608
Record Dates: First submitted 2025-12-15; First posted 2025-12-29 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Primary Dysmenorrhea
Keywords: Pilates exercises; Aerobic exercises
MeSH Terms: interventions — Exercise Movement Techniques; Exercise

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: Pilates exercise group or Aerobic exercise group. Each group will follow a supervised 8week exercise program."
Masking Description: Participants and instructors are not blinded.
  Inclusion Criteria:
  1. Females with Primary dysmenorrhea
  2. Age between 18 to 25 years
  3. Having regular menstrual cycle of 28 - 35 days
  4. Individual with BMI 18.5 to 24.9 kg/m2
  Exclusion Criteria:
  1. Acute or chronic pelvic pathology
  2. Subjects having any history of regular exercises 3days/week [daily average 30-45 min]
  3. Attending physical activity like swimming, running or fitness center
  4. Who cannot perform exercise
  5. Not willing to participate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilates exercises (Experimental): Patients will receive Pilates exercise, the exercise program was repeated 3 times 8 weeks 30 minute for each leg in session. Focused on core strengthening, flexibility, and breathing exercises to alleviate menstrual pain."
  Interventions: Behavioral: Pilates exercises
- Aerobic exercises (Active Comparator): Patients will receive aerobic exercise, the exercise program was repeated 3 times 8 weeks 40minute for each session. Including walk-ing and treadmill
  Interventions: Behavioral: Aerobic exercises

INTERVENTIONS:
Behavioral: Pilates exercises — Patients will receive Pilates exercise, the exercise program was repeated 3 times 8 weeks 30 minute for each leg in session. focuses on core strengthening, flexibility, and breathing techniques designed to reduce menstrual pain and improve overall physical well-being.
  Arms: Pilates exercises
Behavioral: Aerobic exercises — Patients will receive aerobic exercise, the exercise program was repeated 3 times 8 weeks 40minute for each session. Including walk-ing and treadmill
  Arms: Aerobic exercises

SUMMARY:
Comparison between Pilates exercises and aerobic exercises in primary dysmenorrhea

DETAILED DESCRIPTION:
Primary dysmenorrhea is a common gynecological condition among young women and is characterized by painful menstrual cramps that may interfere with daily activities and quality of life. Non-pharmacological interventions, particularly therapeutic exercises, have been recommended as safe and effective approaches for managing menstrual pain. Among these interventions, Pilates exercises and aerobic exercises are widely used; however, comparative evidence regarding their relative effectiveness remains limited.

This study is designed as a comparative interventional trial to evaluate and compare the effects of Pilates exercises versus aerobic exercises on pain severity and quality of life in females with primary dysmenorrhea. Eligible participants will be allocated into two intervention groups.

Participants in Group A will undergo a structured Pilates exercise program conducted three sessions per week for eight weeks. Each session will include controlled movements focusing on core stability, flexibility, breathing control, and muscle strengthening, with a total session duration of approximately 30 minutes.

Participants in Group B will receive a supervised aerobic exercise program performed three sessions per week for eight weeks. The aerobic sessions will consist of rhythmic and continuous movements designed to improve cardiovascular endurance, with each session lasting approximately 40 minutes.

Both interventions will be delivered under standardized conditions, and participants will be instructed to maintain their usual daily activities throughout the study period. Assessments will be conducted before the start of the intervention and after completion of the eight-week exercise program to evaluate changes in menstrual pain severity and quality of life.

The findings of this study aim to provide evidence regarding the comparative effectiveness of Pilates and aerobic exercises in the management of primary dysmenorrhea and to support the selection of appropriate exercise-based interventions for improving pain and quality of life in affected women.

ELIGIBILITY:
Inclusion Criteria:

* Females diagnosed with primary dysmenorrhea
* Age between 18 and 25 years
* Regular menstrual cycle (28-35 days)
* Body mass index (BMI) between 18.5 and 24.9 kg/m²

Exclusion Criteria:

* Presence of any acute or chronic pelvic pathology
* History of regular exercise participation (≥3 days per week, average 30-45 minutes per day)
* Participation in structured physical activities such as swimming, running, or fitness center training
* Inability to perform exercise
* Unwillingness to participate in the study

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-02-10 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
menstrual pain severity | 8 week
  Pain intensity will be measured using the Visual Analog Scale (VAS) atbaseline and after 8 weeks of Pilates or aerobic exercises.low score zero pain and high score 10 worst pain imaginable

SECONDARY OUTCOMES:
Change quality of life | 8weeks
  Short form health survey (SF-12) It was used for assessment of quality of life for aerobic and Pilates before and after treatment.
  higher scores indicating better health, typically on a 0-100 scale where 50 is the average (standardized). A high score (above 50) means better-than-average health, while a low score (below 50) suggests below-average health.

OTHER OUTCOMES:
The Verbal Multidimensional Scoring System (VMSS) | 8weeks
  Assessment include the need for analgesics, systemic symptoms, and ability to work
  , typically scoring from 0 (no pain) to 3 (severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Delta university, Faculty of Physical Therapy, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: No
The study involves a small number of participants, and there is no plan to share individual participant data to ensure privacy and confidentiality.